CLINICAL TRIAL: NCT03326206
Title: Evaluating the Navajo Community Outreach and Patient Empowerment (COPE) Program
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Eastern Research Group, Inc. (Unknown)
Responsible Party: Principal Investigator, Sonya Sunhi Shin, Associate Physician, Brigham and Women's Hospital
Other Study IDs: AD-1304-6566
Record Dates: First submitted 2017-10-24; First posted 2017-10-31 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus; Metabolic Syndrome; Hypertension; Chronic Disease
Keywords: Navajo; Community Health Workers; Community Health Representatives; Tribal health systems; American Indian; Rural; Health disparities
MeSH Terms: conditions — Diabetes Mellitus; Metabolic Syndrome; Hypertension; Chronic Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPE participants: Individuals living with diabetes seen at a study site who were enrolled in the COPE programmatic intervention during the study period. Participation in COPE consists of receiving home visits by a Navajo Community Health Representative (CHR) once or twice a month for a period of at least 12 months. CHRs use structured patient coaching materials to support behavior change. CHRs also check vital signs, monitor blood glucose levels through finger sticks, and facilitate access to appointments and medical refills. CHRs communicate regularly with providers through electronic health record documentation and case management rounds. In-person or telephone communication is be used to address acute issues that may arise.
- Non-COPE participants: Individuals living with diabetes seen at a study site, did not participate in the COPE programmatic intervention, and had comparable baseline characteristics.

SUMMARY:
Since 2009, a programmatic community-based strategy (COPE) has been implemented to address health disparities among Navajo individuals living with multiple chronic conditions. COPE (Community Outreach and Patient Empowerment) targets individual, family, and health system-level factors through four activities: 1) coordination between community health representatives (CHRs) and Indian Health Service providers; 2) CHR competency with standardized training; 3) a culturally-sensitive health promotion curriculum for patients and families; and 4) strong CHR supervision.

COPE has been implemented throughout Navajo Nation. Enrollment is programmatic; in other words, the decision to enroll a patient in COPE occurs independently of whether the patient is in this study. Participants receive the COPE intervention in the same manner and intensity, whether they are included in this observational study or not.

The main goal of this observational research is to understand if COPE improves the lives of participating community members. The Primary Aim is to assess the impact of the COPE Project on changes in HbA1c and other CVD risk factors. Hypothesis: Patients enrolled in the COPE program will experience a reduction in HbA1c compared to the control group. Secondary aims are: 1) To understand if COPE improves patients' own self-reported outcomes. Hypothesis: COPE patients will report better health compared with their own baseline at 12 months. 2) To Identify factors associated with increased effectiveness of the COPE Project at the individual, community, and health system level using a mixed-model approach. 3) To understand diverse stakeholder perspectives on COPE impact and value among CHRs, providers and the health care system. Hypothesis: Compared with baseline, CHRs will report greater empowerment in their work, providers will report greater confidence in CHRs.

The observational cohort will be comprised of individuals with diabetes receiving care at one of the participating health facilities. Cases include individuals participating in the COPE intervention; controls are non-COPE participants identified within the same hospital and matched based on similar baseline characteristics. Study findings will improve clinical and patient-decision making and the health of marginalized AI/ANs by informing policies to promote CHR interventions in rural and underserved communities.

DETAILED DESCRIPTION:
Study population: The study will take place on the Navajo Reservation and within Navajo Area IHS clinical facilities. The Navajo Reservation covers over 27,000 square miles in rural New Mexico and Arizona. The proposed evaluation will occur at the six sites, including two which are currently implementing COPE as well as four sites which will implement COPE in the next two years. The health care centers included in this evaluation represent a mix of federally and tribally operated programs and together provide care for over 200,000 individuals. All sites use a common suite of software applications to record electronic health care data: the IHS RPMS (Resource Patient Management System).

Study Design: The research is aligned with PCORI's definition of patient-centered research by answering questions that will allow patients and other stakeholders to make informed health care decisions. This will be completed by incorporating patient input at all stages; comparatively assessing the benefits and weaknesses of COPE; capturing the "voice" of stakeholders through qualitative methods; choosing outcomes that have been cited as relevant to patients' own priorities and decision-making; and studying cross-site variation to capture individual and community factors associated with impact. The study will address the following questions:

1. Do clinical outcomes (hemoglobin A1c, blood pressure, cholesterol, and body mass index) improve more among COPE participants, compared with similar patients who do not participate in COPE?
2. Do COPE patients experience improvements in self-rated overall health, quality of life, empowerment and satisfaction compared with similar patients who do not participate in COPE?
3. As COPE is implemented in six different service units across the Navajo Nation, can we identify any factors among patients, CHRs, and hospitals that are "key ingredients" for COPE to be effective?
4. Does COPE benefit the health system and population served from diverse stakeholder perspectives including CHRs, providers, and the local health care delivery system?

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes
* Treated at a participating IHS facility corresponding to their home residence

Exclusion Criteria:

* Not seen in one of the six participating clinical sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals receiving care at a Navajo Area Indian Health Service facility, living with diabetes
Sampling Method: Non-Probability Sample
Enrollment: 28813 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonya S Shin, MD MPH, Principal Investigator — Brigham and Women's Hospital
Locations (6):
- United States (6):
  - Chinle Comprehensive Health Care Facility, Chinle, Arizona
  - Tsehootsooi Medical Center, Fort Defiance, Arizona
  - Kayenta Health Center, Kayenta, Arizona
  - Crownpoint Health Center Facility, Crownpoint, New Mexico
  - Gallup Indian Medical Center, Gallup, New Mexico
  - Northern Navajo Medical Center, Shiprock, New Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Franz C, Atwood S, Orav EJ, Curley C, Brown C, Trevisi L, Nelson AK, Begay MG, Shin S. Community-based outreach associated with increased health utilization among Navajo individuals living with diabetes: a matched cohort study. BMC Health Serv Res. 2020 May 25;20(1):460. doi: 10.1186/s12913-020-05231-4. PMID 32450874
- [Derived] Brown C, Lalla A, Curley C, King C, Muskett O, Salt S, Ray K, Begay MG, Nelson AK, Shin S. Community-clinic linkages: qualitative provider perspectives on partnering with community health representatives in Navajo Nation. BMJ Open. 2020 Feb 12;10(2):e031794. doi: 10.1136/bmjopen-2019-031794. PMID 32054623
- [Derived] Lalla A, Salt S, Schrier E, Brown C, Curley C, Muskett O, Begay MG, Shirley L, Clark C, Singer J, Shin S, Nelson AK. Qualitative evaluation of a community health representative program on patient experiences in Navajo Nation. BMC Health Serv Res. 2020 Jan 8;20(1):24. doi: 10.1186/s12913-019-4839-x. PMID 31914997
- [Derived] Trevisi L, Orav JE, Atwood S, Brown C, Curley C, King C, Muskett O, Sehn H, Nelson KA, Begay MG, Shin SS. Integrating community health representatives with health care systems: clinical outcomes among individuals with diabetes in Navajo Nation. Int J Equity Health. 2019 Nov 27;18(1):183. doi: 10.1186/s12939-019-1097-9. PMID 31771603

RESULTS

PARTICIPANT FLOW:
Recruitment Details: COPE participants are recruited to the program as part of routine care. Providers and CHRs identify individuals with uncontrolled chronic diseases, and invite them to participate in the program. Recruitment is programmatic, and not under research auspices.
Groups:
- COPE participants: Individuals with diabetes seen at a study site and enrolled in COPE programmatic intervention during the study period. Participation in COPE consists of receiving home visits by a Navajo Community Health Representative (CHR) once or twice a month for a period of at least 12 months. CHRs deliver structured health coaching, monitor vital signs and blood glucose levels, facilitate access to appointments and medication refills, and communicate with providers to address acute issues that may arise.
- Non-COPE participants: Individuals living with diabetes seen at a study site, did not participate in the COPE programmatic intervention, and had comparable baseline characteristics .
Period: Overall Study - 24 months
Arm/Group | COPE participants | Non-COPE participants
Started | 241 (COPE participants who were identified in study database) | 28572 (Non-COPE participants who were identified in the study database (routine electronic health records))
Completed | 173 (Observational cohort who had data available and able to be matched) | 2880 (Observational cohort who had data available and able to be matched)
Not Completed | 68 | 25692
Not completed — Unable to match cases with controls | 17 | 22721
Not completed — Death | 8 | 92
Not completed — Observational data not available | 43 | 2879
Period: 12 months
Arm/Group | COPE participants | Non-COPE participants
Started | 241 | 28572
Completed | 173 | 2880
Not Completed | 68 | 25692
Not completed — Unable to match cases with controls | 17 | 22721
Not completed — Death | 2 | 50
Not completed — Observational data not available | 49 | 2921

BASELINE CHARACTERISTICS:
Population: The numbers for results differ from those of participant flow because the n for each baseline characteristic depended on data available from health record abstractions.
Groups:
- Total: Total of all reporting groups
Arm/Group | COPE Participants | Non-COPE Participants | Total
Number analyzed (Participants) | 173 | 2880 | 3053
Age, Customized [Count of Participants; unit: Participants]
  18-24 years old | 0 | 0 | 0
  25-40 years old | 7 | 46 | 53
  41-55 years old | 33 | 610 | 643
  56-70 years old | 74 | 1436 | 1510
  71-85 years old | 54 | 764 | 818
  > 85 years old | 5 | 24 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 1979 | 2087
  Male | 65 | 901 | 966
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian / Alaska Native | 173 | 2880 | 3053
  Other | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Navajo Area Indian Health Services | 173 | 2880 | 3053
  United States: Other | 0 | 0 | 0
Preferred language [Count of Participants; unit: Participants] — Population: Data missing on variable in observational database
  Participants
    number analyzed (Participants) | 172 | 2878 | 3050
    Navajo or other Native American language | 100 | 1178 | 1278
    English | 72 | 1700 | 1772
Primary Care Physician [Count of Participants; unit: Participants]
  Primary Care Provider assigned | 146 | 2577 | 2723
  No Primary Care Provider assigned | 27 | 303 | 330
Essential hypertension [Count of Participants; unit: Participants] — Population: Data missing on variable in observational database
  Participants
    number analyzed (Participants) | 173 | 2875 | 3048
    Yes | 113 | 1966 | 2079
    No | 60 | 909 | 969
Major Depressive Disorder [Count of Participants; unit: Participants] — Population: Data missing on variable in observational database
  Participants
    number analyzed (Participants) | 173 | 2875 | 3048
    Yes | 25 | 282 | 307
    No | 148 | 2593 | 2741
Major cardiovascular disease [Count of Participants; unit: Participants] — Population: Data missing on variable in observational database
  Participants
    number analyzed (Participants) | 173 | 2875 | 3048
    Yes | 123 | 2050 | 2173
    No | 50 | 825 | 875
Dyslipidemia [Count of Participants; unit: Participants] — Population: Data missing on variable in observational database
  Participants
    number analyzed (Participants) | 173 | 2875 | 3048
    Yes | 80 | 1688 | 1768
    No | 93 | 1187 | 1280
Alcohol Use Disorder [Count of Participants; unit: Participants] — Population: Data missing on variable in observational database
  Participants
    number analyzed (Participants) | 173 | 2875 | 3048
    Yes | 11 | 77 | 88
    No | 162 | 2798 | 2960

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage of Glycated Hemoglobin (HbA1c)
Description: Change in Hemoglobin A1c measured at 24 months, compared with baseline
Time Frame: 24 months
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | COPE participants | Non-COPE participants
Number analyzed (Participants) | 173 | 2880
percent | -0.49 [-0.62 to -0.37] | 0.13 [0.10 to 0.17]
Statistical Analysis 1: Comparison: COPE participants vs Non-COPE participants; Mixed linear regression models were performed to assess differences over time for continuous variables, comparing COPE versus control groups. The models included a random effect for patients to account for within-patient correlation over time in the outcome measures and a random effect for the primary health facility, to account for within-site correlation. In the sensitivity analyses we also adjusted the models for the random effect of matching groups; Test type: Superiority; p < 0.0001, Regression, Linear — A priori threshold for statistical significance < 0.05; Mixed linear regression

2. Secondary Outcome: Change in Systolic Blood Pressure
Description: Changes in systolic blood pressure at 24 months, compared with baseline
Time Frame: 24 months
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | COPE participants | Non-COPE participants
Number analyzed (Participants) | 173 | 2880
mmHg | 1.43 [0.67 to 2.18] | 0.28 [0.06 to 0.50]
Statistical Analysis 1: Comparison: COPE participants vs Non-COPE participants; Test type: Superiority; p = 0.004, Regression, Linear — a priori threshold for significance p<0.05; Mixed linear regression as described in primary endpoint

3. Secondary Outcome: Change in Low-density Lipoprotein
Description: Change in low density lipoprotein at 24 months, compared with baseline
Time Frame: 24 months
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | COPE participants | Non-COPE participants
Number analyzed (Participants) | 173 | 2880
mg/dl | -8.04 [-11.88 to -4.20] | -3.21 [-4.17 to -2.24]
Statistical Analysis 1: Comparison: COPE participants vs Non-COPE participants; Test type: Superiority; p = 0.02, Regression, Linear — a priori threshold for significant p<0.05; Mixed linear regression as described in primary endpoint

4. Secondary Outcome: Change in Body Mass Index
Description: change in body mass index at 24 months, compared with baseline
Time Frame: 24 months
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | COPE participants | Non-COPE participants
Number analyzed (Participants) | 173 | 2880
kg/m^2 | -0.25 [-0.51 to 0.01] | -0.26 [-0.34 to -0.18]
Statistical Analysis 1: Comparison: COPE participants vs Non-COPE participants; Test type: Superiority; p = 0.93, Regression, Linear — a priori threshold for significance p<0.05; Mixed linear regression model as described for primary endpoint

5. Secondary Outcome: Change in Primary Outpatient Services
Description: Primary outpatient encounters are identified using the Resource Patient Management System (RPMS) clinic variable. It is notable that the clinic variable includes types of health utilization that are not limited to clinic visits, e.g. inpatient, emergency primary, specialty, dental, counseling/behavioral care. Each clinic visit reported in RPMS is counted as one utilization incident for the purposes of this analysis.
Time Frame: 24 months
Measure: Least Squares Mean (95% Confidence Interval); unit: number of visits per quarter post enroll
Arm/Group | COPE participants | Non-COPE participants
Number analyzed (Participants) | 173 | 2885
number of visits per quarter post enroll | 1.0750 [0.9618 to 1.2016] | 0.9224 [0.8952 to 0.9505]
Statistical Analysis 1: Comparison: COPE participants vs Non-COPE participants; Generalized linear mixed regression models were used for count outcomes (SAS 9.3: PROC GLIMMIX) to estimate change in health care visits by COPE pts relative to non-COPE pts. Random effects accounted for within-site correlation at service units. Adjusted for covariates: age, gender, language, primary care physician, and diagnoses: essential hypertension, major depression disorder, alcohol abuse, major cardiovascular disease, and dyslipidemia; Test type: Superiority; p = 0.0091, Regression, Linear — Primary result is coefficient on post intervention change in visits by COPE pts relative to controls: if significant and >0, COPE visits have increased relative to controls; if significant and <0, COPE visits have decreased relative to controls

6. Secondary Outcome: Change in Specialty Outpatient Services
Description: Specialty outpatient encounters are identified using the Resource Patient Management System (RPMS) clinic variable. It is notable that the clinic variable includes types of health utilization that are not limited to clinic visits, e.g. inpatient, emergency primary, specialty, dental, counseling/behavioral care. Each clinic visit reported in RPMS is counted as one utilization incident for the purposes of this analysis.
Time Frame: 24 months
Measure: Least Squares Mean (95% Confidence Interval); unit: number of visits per quarter post enroll
Arm/Group | COPE participants | Non-COPE participants
Number analyzed (Participants) | 173 | 2885
number of visits per quarter post enroll | 0.8856 [0.7720 to 1.0160] | 0.6838 [0.6610 to 0.7074]
Statistical Analysis 1: Comparison: COPE participants vs Non-COPE participants; As described for primary outpatient services; Test type: Superiority; p = 0.0003, Regression, Linear

7. Secondary Outcome: Change in Emergency Services
Description: Emergency encounters are identified using the Resource Patient Management System (RPMS) clinic variable. It is notable that the clinic variable includes types of health utilization that are not limited to clinic visits, e.g. inpatient, emergency primary, specialty, dental, counseling/behavioral care. Each clinic visit reported in RPMS is counted as one utilization incident for the purposes of this analysis.
Time Frame: 24 months
Measure: Least Squares Mean (95% Confidence Interval); unit: number of visits per quarter post enroll
Arm/Group | COPE participants | Non-COPE participants
Number analyzed (Participants) | 173 | 2885
number of visits per quarter post enroll | 0.2755 [0.2306 to 0.3290] | 0.2559 [0.2448 to 0.2674]
Statistical Analysis 1: Comparison: COPE participants vs Non-COPE participants; as described for primary outpatient services; Test type: Superiority; p = 0.4296, Regression, Linear

8. Secondary Outcome: Change in Counseling / Behavioral Services
Description: Counseling / behavioral encounters are identified using the Resource Patient Management System (RPMS) clinic variable. It is notable that the clinic variable includes types of health utilization that are not limited to clinic visits, e.g. inpatient, emergency primary, specialty, dental, counseling/behavioral care. Each "clinic visit" reported in RPMS is counted as one utilization incident for the purposes of this analysis.
Time Frame: 24 months
Measure: Least Squares Mean (95% Confidence Interval); unit: number of visits per quarter post enroll
Arm/Group | COPE participants | Non-COPE participants
Number analyzed (Participants) | 173 | 2885
number of visits per quarter post enroll | 0.2590 [0.2164 to 0.3101] | 0.1432 [0.1363 to 0.1504]
Statistical Analysis 1: Comparison: COPE participants vs Non-COPE participants; As described for primary outpatient services; Test type: Superiority; p < 0.0001, Regression, Linear

9. Secondary Outcome: Change in Laboratory Services
Description: Laboratory encounters are identified using the Resource Patient Management System (RPMS) clinic variable. It is notable that the clinic variable includes types of health utilization that are not limited to clinic visits, e.g. inpatient, emergency primary, specialty, dental, counseling/behavioral care. Each "clinic visit" reported in RPMS is counted as one utilization incident for the purposes of this analysis.
Time Frame: 24 months
Measure: Least Squares Mean (95% Confidence Interval); unit: number of visits per quarter post enroll
Arm/Group | COPE participants | Non-COPE participants
Number analyzed (Participants) | 173 | 2885
number of visits per quarter post enroll | 0.3510 [0.2838 to 0.4341] | 0.2798 [0.2650 to 0.2955]
Statistical Analysis 1: Comparison: COPE participants vs Non-COPE participants; Test type: Superiority; p = 0.0431, Regression, Linear

10. Secondary Outcome: Change in Radiology Services
Description: Radiology encounters are identified using the Resource Patient Management System (RPMS) clinic variable. It is notable that the clinic variable includes types of health utilization that are not limited to clinic visits, e.g. inpatient, emergency primary, specialty, dental, counseling/behavioral care. Each "clinic visit" reported in RPMS is counted as one utilization incident for the purposes of this analysis.
Time Frame: 24 months
Measure: Least Squares Mean (95% Confidence Interval); unit: encounters per patient per quarter
Arm/Group | COPE participants | Non-COPE participants
Number analyzed (Participants) | 173 | 2885
encounters per patient per quarter | 0.0304 [0.0222 to 0.0416] | 0.0220 [0.0202 to 0.0240]
Statistical Analysis 1: Comparison: COPE participants vs Non-COPE participants; Test type: Superiority; p = 0.0516, Regression, Linear

11. Secondary Outcome: Change in Pharmacy Services
Description: Pharmacy encounters are identified using the Resource Patient Management System (RPMS) clinic variable. It is notable that the clinic variable includes types of health utilization that are not limited to clinic visits, e.g. inpatient, emergency primary, specialty, dental, counseling/behavioral care. Each "clinic visit" reported in RPMS is counted as one utilization incident for the purposes of this analysis.
Time Frame: 24 months
Measure: Least Squares Mean (95% Confidence Interval); unit: number of visits per quarter post enroll
Arm/Group | COPE participants | Non-COPE participants
Number analyzed (Participants) | 173 | 2885
number of visits per quarter post enroll | 0.5477 [0.4816 to 0.6229] | 0.5146 [0.4977 to 0.5321]
Statistical Analysis 1: Comparison: COPE participants vs Non-COPE participants; Test type: Superiority; p = 0.3582, Regression, Linear

12. Secondary Outcome: Change in Inpatient Services
Description: For inpatient services, the primary data point is the presence of a DRG code indicating the patient was hospitalized. However, we also included clinic listings for labor and delivery and for observation as inpatient utilization.
Time Frame: 24 months
Measure: Least Squares Mean (95% Confidence Interval); unit: number of visits per quarter post enroll
Arm/Group | COPE participants | Non-COPE participants
Number analyzed (Participants) | 173 | 2885
number of visits per quarter post enroll | 0.1869 [0.1436 to 0.2433] | 0.1592 [0.1491 to 0.1699]
Statistical Analysis 1: Comparison: COPE participants vs Non-COPE participants; Test type: Superiority; p = 0.2461, Regression, Linear

13. Secondary Outcome: Change in Dental Encounters
Description: Dental encounters are identified using the Resource Patient Management System (RPMS) clinic variable. It is notable that the clinic variable includes types of health utilization that are not limited to clinic visits, e.g. inpatient, emergency primary, specialty, dental, counseling/behavioral care. Each clinic visit reported in RPMS is counted as one utilization incident for the purposes of this analysis.
Time Frame: 24 months
Measure: Least Squares Mean (95% Confidence Interval); unit: number of visits per quarter post enroll
Groups:
- COPE participants: Individuals living with diabetes seen at a study site who were enrolled in the COPE programmatic intervention during the study period.
Arm/Group | COPE participants | Non-COPE participants
Number analyzed (Participants) | 173 | 2885
number of visits per quarter post enroll | 0.1119 [0.0875 to 0.1429] | 0.1422 [0.1344 to 0.1505]
Statistical Analysis 1: Comparison: COPE participants vs Non-COPE participants; Test type: Superiority; p = 0.0613, Regression, Linear

14. Secondary Outcome: Change in Community Encounters
Description: Community encounters are identified using the Resource Patient Management System (RPMS) clinic variable. Community Encounters may include public health nursing and community health representative visits; however, not all community encounters (e.g. visits by Community Health Representatives in clinics where Community Health Representatives do not document their visits on the RPMS system) may be represented in this database
Time Frame: 24 months
Measure: Least Squares Mean (95% Confidence Interval); unit: number of visits per quarter post enroll
Groups:
- COPE participants: Individuals with diabetes seen at a study site and enrolled in COPE programmatic intervention during the study period.
Arm/Group | COPE participants | Non-COPE participants
Number analyzed (Participants) | 173 | 2885
number of visits per quarter post enroll | 0.1160 [0.0900 to 0.1497] | 0.0189 [0.0171 to 0.0207]
Statistical Analysis 1: Comparison: COPE participants vs Non-COPE participants; Test type: Superiority; p < 0.0001, Regression, Linear

15. Other Pre Specified Outcome: Patient-reported Good Health
Description: Health status is assessed by three questions using a 5-point scale response to the General Health question from the Short Form 12 survey: "Would you say that in general your health is…" "Compared to your health a year ago, would you say your health is" and "Compared to other people your age, would you say your health is" (Excellent=5, Very Good=4, Good=3, Fair=2, Poor=1), where higher values are more favorable.
  Binary outcome of Good Health includes "Excellent," "Very good" and "Good" as yes, other responses as no.
Time Frame: 12 months
Population: For this outcome, only pre-post analysis was collected among a subset of COPE participants (rather than COPE v. non-COPE arms)
Measure: Count of Participants; unit: Participants
Groups:
- COPE participants - baseline: Survey data administered to patients at the time of enrollment into the COPE Program
- COPE participants - 12 months: Surveys administered to patients after 1 year of participation in the COPE program
Arm/Group | COPE participants - baseline | COPE participants - 12 months
Number analyzed (Participants) | 22 | 22
Participants
  Good health: Yes | 15 | 12
  Good health: No | 7 | 10
  Good health compared to a year ago: Yes | 13 | 18
  Good health compared to a year ago: No | 9 | 4
  Good health compared to other people your age: Yes | 13 | 18
  Good health compared to other people your age: No | 9 | 4
Statistical Analysis 1: Comparison: COPE participants - baseline vs COPE participants - 12 months; Test type: Superiority; p = 0.54, Fisher Exact

16. Other Pre Specified Outcome: Patient-reported Sense of Control
Description: Sense of control is assessed using a 4-point scale response to the question "Do you feel you are in control of your health?" (Always Never=1, Rarely=2, Sometimes=3, Almost Always=4) with a higher value representing a favorable outcome. Binary outcome derived by including "Almost Always" in "Yes" and "Always never," "Rarely" and "Sometimes" in "No"
Time Frame: 12 months
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | COPE participants - baseline | COPE participants - 12 months
Number analyzed (Participants) | 22 | 22
Participants
  Yes | 7 | 10
  No | 15 | 12
Statistical Analysis 1: Comparison: COPE participants - baseline vs COPE participants - 12 months; Test type: Superiority; p = 0.19, Chi-squared — P-value corresponds to patient-reported health compared to a year ago and compared to others their age

17. Other Pre Specified Outcome: Patient-reported Ability to Cope
Description: Coping will be assessed using a 4-point scale response to two questions "how often have you found that you couldn't cope with all the things that you had to do to?" (Always Never=4, Rarely=3, Sometimes=2, Almost Always=1) and "In the last month, how often have you been upset because of something that happened unexpectedly?" (Always Never=4, Rarely=3, Sometimes=2, Almost Always=1) with a higher value representing a favorable outcome. Binary variables derived by grouping "Always never" and "Rarely" as "Yes" and all others responses as "No"
Time Frame: 12 months
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | COPE participants - baseline | COPE participants - 12 months
Number analyzed (Participants) | 22 | 22
Participants
  Able to cope with all the things you had to do: Yes | 6 | 14
  Able to cope with all the things you had to do: No | 16 | 8
  Able to cope with unexpected negative events: Yes | 2 | 12
  Able to cope with unexpected negative events: No | 20 | 10
Statistical Analysis 1: Comparison: COPE participants - baseline vs COPE participants - 12 months; Test type: Superiority; p = 0.0028, Fisher Exact — P value corresponds with Ability to cope with negative life events

ADVERSE EVENTS:
Time Frame: 24 months
Description: Because this study was an observational, prospective study, adverse events are reported based on routine clinical data during the study period: 1) all-cause mortality; 2) serious adverse events defined as incident cardiovascular disease; 3) non serious adverse events were not collected
Arm/Group | COPE participants | Non-COPE participants
All-Cause Mortality (participants affected / at risk) | 8/173 | 92/2885
Serious Adverse Events (participants affected / at risk) | 2/173 | 3/2885
Other Adverse Events (participants affected / at risk) | 54/173 | 493/2885
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COPE participants (N=173) | Non-COPE participants (N=2885)
Incident CVD (Cardiac disorders) | 2 (2) | 3 (3) — acute myocardial infarction, coronary artery bypass surgery, coronary angioplasty, peripheral arterial disease, abdominal aortic aneurysm, carotid artery disease, cerebrovascular disease
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COPE participants (N=173) | Non-COPE participants (N=2885)
Inpatient hospitalization (Endocrine disorders) | 54 (145) | 493 (790) — Any inpatient hospitalization event, due to any cause.

LIMITATIONS AND CAVEATS:
This is an observational study using routine clinical data for endpoints other than patient-reported outcomes. Therefore, the participant flow and adverse event reporting did not conform to clinical trial protocols. For patient-reported outcomes, we used mixed methods (including pre-post surveys among a sub-set of COPE participants and qualitative interviews) but did not collect or compare data from a control arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No